CLINICAL TRIAL: NCT02440412
Title: Effects of a Single Session of Massage Therapy in Salivary Cortisol Levels in Asymptomatic Persons With Administrative Tasks and / or Office Work.
Brief Title: Effect of Massage Therapy in Cortisol Level
Acronym: MTCL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Rodrigo Antonio Rojo Castro, Academic Of Department of Physical Therapy, University of Chile
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Kine015
Record Dates: First submitted 2015-05-01; First posted 2015-05-12 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Asymptomatic State
Keywords: Massage; Stress; salivary cortisol
MeSH Terms: conditions — Asymptomatic Diseases | interventions — Massage; RE1-silencing transcription factor; Supine Position

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Massage Therapy (Experimental): A 45 minutes massage therapy (manual) standardized session, based in Swedish techniques.
  Interventions: Other: Massage Therapy
- Rest condition (Placebo Comparator): 45 minutes of rest in supine position, listening music with headphones, and warm condition.
  Interventions: Other: Rest in supine
- Control (No Intervention): Normal working condition, as a office workers (secretaries and managements employees)

INTERVENTIONS:
Other: Massage Therapy — It's a Physical Therapy manual procedure, based in Swedish technique, and applied in a standirzed way for all participants (stroke, kneading, pressure).
  Arms: Massage Therapy
Other: Rest in supine — It's only rest, in a clinic stretcher, with warm ambient temperature, and listening relaxing music with headphones.
  Arms: Rest condition

SUMMARY:
This study evaluates the effect of a single session of Massage Therapy in salivary cortisol level. All participants were assessed on three conditions: Massage session, rest in supine position listening music, and under normal working conditions. The hypothesis of the investigators is that the effect of the massage action in reduction of cortisol is superior to only rest.

DETAILED DESCRIPTION:
Several studies have postulated that one of the physiological markers of the effect of massage therapy is to reduce the level of cortisol, the "stress hormone". However it is not clear whether the effect is due to the manual action on the skin, or only by the relaxation induced rest. Therefore the variation of salivary cortisol in both conditions, and also in everyday working conditions was compared. Cortisol has a circadian cycle, with a maximum value upon awakening, which decreases during the morning; therefore a sample of saliva (in Salivette tube) it was collected in the three experimental conditions at the same hour time in the morning: 8:45(after intervention), and 9:30 and 10.30 (both, before).

ELIGIBILITY:
Inclusion Criteria:

* Office/administrative workers of Faculty of Medicine, University of Chile.

Exclusion Criteria:

* Musculoskeletal disease or injury in spine.
* Body Mass Index over 35.
* Smoking (over three cigars at day)
* Depression.
* Pregnancy
* Corticosteroid treatment.
* Skin wound or disease.
* Intolerance to the prone position.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-07; Primary Completion 2014-11 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change of Salivary Cortisol Level | All participants were measured in three different condition, one week apart one each other. In each condition, three measurements were performed, in the morning
  Data (a saliva sample in a Salivette (r) tube) were collected at: immediately before the intervention and placebo procedure, immediately after and later, one hour after. The control condition (normal working condition) was measured at the same hours (8:45 AM, 9.30 AM and 10.30 AM) in the workplace. After collected, were refrigerated.The three conditions (intervention, placebo and office work) were a week apart. Therefore, each participant had nine measurements. Determining the level of cortisol was performed by ELISA method, after all samples were collected.

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo A Rojo, Msc., Principal Investigator — Physical Therapy Department, University of Chile
Locations (1):
- Faculty of Medicine, University of Chile, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- [Background] Moyer CA, Rounds J, Hannum JW. A meta-analysis of massage therapy research. Psychol Bull. 2004 Jan;130(1):3-18. doi: 10.1037/0033-2909.130.1.3. PMID 14717648
- [Result] Rapaport MH, Schettler P, Bresee C. A preliminary study of the effects of repeated massage on hypothalamic-pituitary-adrenal and immune function in healthy individuals: a study of mechanisms of action and dosage. J Altern Complement Med. 2012 Aug;18(8):789-97. doi: 10.1089/acm.2011.0071. Epub 2012 Jul 9. PMID 22775448
- [Result] Field T, Ironson G, Scafidi F, Nawrocki T, Goncalves A, Burman I, Pickens J, Fox N, Schanberg S, Kuhn C. Massage therapy reduces anxiety and enhances EEG pattern of alertness and math computations. Int J Neurosci. 1996 Sep;86(3-4):197-205. doi: 10.3109/00207459608986710. PMID 8884390
- [Result] Lindgren L, Rundgren S, Winso O, Lehtipalo S, Wiklund U, Karlsson M, Stenlund H, Jacobsson C, Brulin C. Physiological responses to touch massage in healthy volunteers. Auton Neurosci. 2010 Dec 8;158(1-2):105-10. doi: 10.1016/j.autneu.2010.06.011. PMID 20638912
- [Result] Arroyo-Morales M, Olea N, Ruiz C, del Castilo Jde D, Martinez M, Lorenzo C, Diaz-Rodriguez L. Massage after exercise--responses of immunologic and endocrine markers: a randomized single-blind placebo-controlled study. J Strength Cond Res. 2009 Mar;23(2):638-44. doi: 10.1519/JSC.0b013e318196b6a6. PMID 19197204
- [Result] Lovas J. The effects of massage therapy on the human immune response in healthy adults. J Bodyw Mov Ther. 2002; 143-150
- [Result] Moyer CA, Seefeldt L, Mann ES, Jackley LM. Does massage therapy reduce cortisol? A comprehensive quantitative review. J Bodyw Mov Ther. 2011 Jan;15(1):3-14. doi: 10.1016/j.jbmt.2010.06.001. Epub 2010 Jul 2. PMID 21147413
- [Result] Field T, Diego M, Hernandez-Rief M. Massage therapy research. Developmental Review. 2007; 27: 75-8
- [Result] Field T, Diego M, Cullen C, Hernandez-Reif M, Sunshine W, Douglas S. Fibromyalgia pain and substance P decrease and sleep improves after massage therapy. J Clin Rheumatol. 2002 Apr;8(2):72-6. doi: 10.1097/00124743-200204000-00002. PMID 17041326
- [Result] Field T, Hernandez-Reif M, Diego M, Schanberg S, Kuhn C. Cortisol decreases and serotonin and dopamine increase following massage therapy. Int J Neurosci. 2005 Oct;115(10):1397-413. doi: 10.1080/00207450590956459. PMID 16162447
- [Result] Moraska A, Pollini RA, Boulanger K, Brooks MZ, Teitlebaum L. Physiological adjustments to stress measures following massage therapy: a review of the literature. Evid Based Complement Alternat Med. 2010 Dec;7(4):409-18. doi: 10.1093/ecam/nen029. Epub 2008 May 7. PMID 18955340
- [Result] Field T. Massage therapy research review. Complement Ther Clin Pract. 2014 Nov;20(4):224-9. doi: 10.1016/j.ctcp.2014.07.002. Epub 2014 Aug 1. PMID 25172313